CLINICAL TRIAL: NCT04889924
Title: Axillary Lymph Node Dissection Versus Axillary Radiotherapy in Breast Cancer Patients With Positive Sentinel Node After Neoadjuvant Therapy: A Multicenter Randomized Study
Brief Title: ALND vs ART in Positive Sentinel Node After Neoadjuvant Therapy in Breast Cancer
Acronym: ADARNAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR148/21
Record Dates: First submitted 2021-05-05; First posted 2021-05-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Chemotherapy; Sentinel Lymph Node; Axillary Lymph Nodes Dissection; Radiotherapy Side Effect
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries | interventions — Lymph Node Excision

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, multicenter study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axillary radiotherapy without lymphadenectomy (Experimental): Axillary radiotherapy (level I and II) + level III and supraclavicular +/- internal mammary chain without lymphadenectomy
  Interventions: Radiation: Axillary Radiotherapy
- Axillary lymph node dissection (Active Comparator): Axillary lymph node dissection + radiotherapy level III and supraclavicular +/- internal mammary chain
  Interventions: Procedure: Lymphadenectomy

INTERVENTIONS:
Radiation: Axillary Radiotherapy — Axillary radiotherapy without lymphadenectomy (level I and II) + level III and supraclavicular +/- internal mammary chain
  Arms: Axillary radiotherapy without lymphadenectomy
Procedure: Lymphadenectomy — Axillary lymph node dissection + radiotherapy level III and supraclavicular +/- internal mammary chain
  Arms: Axillary lymph node dissection

SUMMARY:
In the case of primary surgery, in patients with sentinel node involvement, it has already been shown that omitting axillary lymph node dissection (ALND), often combining axillary radiotherapy (RT), does not worsen the prognosis and does significantly reduce the appearance of lymphedema. However, patients who have received neoadjuvant systemic treatment cannot benefit from this option, even though in the majority of those who have responded well to treatment, a residual disease in the armpit is low, but there are no studies yet published that supports the possibility of not performing lymphadenectomy.

The primary endpoint is to evaluate wether axillary radiotherapy (ART) presents a lower risk of lymphedema with respect to lymphadenectomy (ALND) in patients with breast cancer who, after neoadjuvant systemic treatment (NST), present the sentinel node affected. Likewise, we will evaluate recurrences and overall survival in both groups. Finally, we will analyze the quality of life of these patients.

DETAILED DESCRIPTION:
A prospective, randomized, open-label, parallel-assigned, multicenter study. The estimated sample size is 820 patients (410 patients in neoadjuvant chemotherapy and 410 in neoadjuvant hormone therapy), over 5 years. Patients will be stratified and analyzed independently according to the neoadjuvant treatment regimen, whether chemotherapy (CT) +/- hormonal therapy (HT).

A pilot phase of the study was carried out with the first 200 patients (Until 1 May 2023), and an interim analysis will also be performed with these first 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* T1-T4 N0/ T0-T4 N1 at diagnosis and subsidiary of neoadjuvant treatment
* Post-CT SLN with ≤2 macrometastasis/micrometastasis or ITCs
* Post-CT axillary response by ultrasound or MRI
* Complete at least 70% of neoadjuvant chemotherapy and 6 months of endocrine treatment.

Exclusion Criteria:

* cN2
* ypN0
* History of breast surgery for ipsilateral cancer in the last 10 years
* History of other cancer in the last 5 years, except squamous carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From date of diagnosis until the date of first documented recurrence or death, wichever came first,assessed up to 5 years
  To assess whether the irradiation of the axilla concerning axillary lymph node dissection is not inferior in disease-free survival, in patients with positive sentinel lymph node (SN) after neoadjuvant systemic treatment.

SECONDARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause, assessed up to 5 years
  To assess whether the irradiation of the axilla concerning axillary lymph node dissection is not inferior in overall survival, in patients with positive sentinel lymph node (SN) after neoadjuvant systemic treatment.
Lymphedema Incidence | From date of surgery until the date of first lynphedema apparition, assessed up to 3 years
  Volume difference between both arms (cm^3) above 10%

CONTACTS AND LOCATIONS:
Overall Officials: Maria Laplana, MDPhD, Principal Investigator — Hospital Clínico y Provincial de Barcelona; Amparo Garcia-Tejedor, MDPhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (58):
- Australia (6):
  - GenesisCare Mater, Sydney, New South Wales
  - GenesisCare North Shore, Sydney, New South Wales
  - GenesisCare Frenchs Forest, Sydney, New South Wales
  - GenesisCare Norwest, Sydney, New South Wales
  - GenesisCare Hurstville, Sydney, New South Wales
  - GenesisCare Campbelltown, Sydney, New South Wales
- Spain (52):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Instituto Catalán de Oncología de Badalona, Badalona, Barcelona
  - Hospital Comarcal Sant Jaume de Calella, Calella, Barcelona
  - Consorci Sanitari Integral, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Instituto Catalán de Oncología- Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Fundación Althaia Manresa, Manresa, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Universitario General de Cataluña, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Mútua Terrassa, Terrassa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital de Viladecans, Viladecans, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Galdakao-Usansolo, Galdakao, Bizkaia
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta De Hierro, Majadahonda, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Ribera Povisa, Vigo, Pontevedra
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Cruz y San Pablo, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de Gerona Doctor Josep Trueta, Girona
  - Institut Catalán de Oncología de Girona, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Infanta Sofía- Fundación de Inv. Biomédica H. Infanta Sofía, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Montecelo, Pontevedra
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital General de Segovia, Segovia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario de Tarragona Juan XXIII, Tarragona
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Recoletas Campo Grande de Valladolid, Valladolid
  - Hospital Universitario de Álava / Txagorritxu, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Tejedor A, Ortega-Exposito C, Salinas S, Luzardo-Gonzalez A, Falo C, Martinez-Perez E, Perez-Montero H, Soler-Monso MT, Bajen MT, Benitez A, Ortega R, Petit A, Guma A, Campos M, Pla MJ, Pernas S, Penafiel J, Yeste C, Gil-Gil M, Guedea F, Ponce J, Laplana M. Axillary lymph node dissection versus radiotherapy in breast cancer with positive sentinel nodes after neoadjuvant therapy (ADARNAT trial). Front Oncol. 2023 Aug 9;13:1184021. doi: 10.3389/fonc.2023.1184021. eCollection 2023. PMID 37621686